CLINICAL TRIAL: NCT02070185
Title: Effect of Energy Density on Liking and on Caloric Adjustment Conditioning After Sweet Beverage Exposure in Children Aged 8-11 y
Brief Title: Effect of Energy Density on Liking and on Caloric Adjustment Conditioning
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut National de Recherche pour l'Agriculture, l'Alimentation et l'Environnement (Other)
Collaborators: European Community (Unknown); Regional Council of Burgundy (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: Energy
Record Dates: First submitted 2014-02-17; First posted 2014-02-25 (Estimated); Last update posted 2014-02-25 (Estimated); Status verified 2014-02

CONDITIONS: Conditioning of Caloric Adjustment and Liking in Children
Keywords: caloric adjustment,liking, flavour nutrient learning, children

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 2 exposures (Experimental): During the conditioning period, the children of this group was exposed only twice to the beverages
  Interventions: Behavioral: 2 exposures arm
- 7 exposures (Experimental): During the conditioning period, children of this group were exposed exposed 7 times to the beverages
  Interventions: Behavioral: 7 exposures arm

INTERVENTIONS:
Behavioral: 2 exposures arm — During this study, children were exposed to 2 flavored sweetened beverages: a high energy version (HE: 150kcal) and a no energy version (NE: 0kcal).
  During a 4-wk conditioning period, children were exposed either 2 times to each beverage.
  After a 3-wk stability period without exposure, children were exposed 3 times to both beverages in which the association between the flavor and the energy density had been switched (4-wk extinction period).
  Arms: 2 exposures
Behavioral: 7 exposures arm — During this study, children were exposed to 2 flavored sweetened beverages: a high energy version (HE: 150kcal) and a no energy version (NE: 0kcal).
  During a 4-wk conditioning period, children were exposed either 7 times to each beverage.
  After a 3-wk stability period without exposure, children were exposed 3 times to both beverages in which the association between the flavor and the energy density had been switched (4-wk extinction period).
  Arms: 7 exposures

SUMMARY:
The main objective is to study, in 8-11 year old children, the influence of energy density conditioning on liking for new flavored beverages and on caloric adjustment after the beverage consumption. The stability of the energy conditioning was evaluated after a period without exposure and after an extinction period during which the energy density of the beverages was changed.

ELIGIBILITY:
Inclusion Criteria:

* regularly ate at the school canteen
* returned signed consent from parents

Exclusion Criteria:

* present health problems, food restrictions or food allergies

Ages: 8 Years to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 45 (Actual)
Dates: Start 2013-03; Primary Completion 2013-03 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Flavored beverages liking and preference before the conditioning period (T0) | Baseline
  Liking and preference measurements for the flavored beverages, before the conditioning period.

SECONDARY OUTCOMES:
Energy adjustment before the conditioning period (T0) | Baseline
  Measure of energy intake at the lunch following the beverage consumption, before the conditioning period

OTHER OUTCOMES:
Energy adjustment after the conditioning period (T1) | T0 + 4 weeks
  Measure of energy intake at the lunch following the beverage consumption, after the 4-week conditioning period
Flavored beverages liking and preference after the conditioning period (T1) | T0 + 4 weeks
  Liking and preference measurements for the new flavored beverages, after the 4-week conditioning period.
Flavored beverages liking and preference after 3 weeks without exposure (T2) | T1 + 3 weeks
  liking and preference measurements of the new flavored beverages, after a period of 3 weeks without exposure (=stability period)
Flavored beverages liking and preference before the extinction period (T3) | T2 +1 week
  Liking and preference measurements of the new flavored beverages before a 4-week- extinction period during which the energy density of the beverages were changed
Energy adjustment before an extinction period (T3) | T2 + 1 week
  Measure of energy intake at the lunch following the beverages consumption,before the 4-week- extinction period, during which the energy density of the beverages were changed.
Energy adjustment after 3 weeks without exposure (T2) | T1 + 3 weeks
  Measure of energy intake at lunch following the beverage consumption, after a period of 3 weeks without exposure
Energy adjustment after the extinction period (T4) | T3 + 4 weeks
  Measure of energy intake at the lunch following the beverages consumption,after the 4-week- extinction period, during which the energy density of the beverages were changed.
Flavored beverages liking and preference before the extinction period (T4) | T3 + 4 weeks
  Liking and preference measurements of the new flavored beverages after the 4-week- extinction period during which the energy density of the beverages were changed

CONTACTS AND LOCATIONS:
Locations (1):
- Centre des Sciences du Goût et de l'Alimentation, Dijon, Bourgogne-Franche-Comté, France

REFERENCES:
- [Derived] Remy E, Divert C, Rousselot J, Brondel L, Issanchou S, Nicklaus S. Impact of energy density on liking for sweet beverages and caloric-adjustment conditioning in children. Am J Clin Nutr. 2014 Oct;100(4):1052-8. doi: 10.3945/ajcn.114.087452. Epub 2014 Aug 13. PMID 25240072